CLINICAL TRIAL: NCT01774253
Title: A Phase II, Open-label, Multi-center Study of Erivedge (Vismodegib) in the Treatment of Pediatric Patients With Refractory Pontine Glioma.
Brief Title: Erivedge (Vismodegib) in the Treatment of Pediatric Patients With Refractory Pontine Glioma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of enrollment and commercial availability of drug
Sponsor: Giselle Sholler (Other)
Collaborators: Phoenix Children's Hospital (Other)
Responsible Party: Sponsor-Investigator, Giselle Sholler, Beat Childhood Cancer Chair, Milton S. Hershey Medical Center
Organization: Milton S. Hershey Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NMTRCPG007
Record Dates: First submitted 2013-01-18; First posted 2013-01-23 (Estimated); Results first posted 2016-10-28 (Estimated); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Pontine Glioma
Keywords: DIPG
MeSH Terms: interventions — HhAntag691

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vismodegib (Experimental): Vismodegib will be dosed at 150mg-300mg orally (max dose: 300mg) once a day on days 1 to 28 of a 28-day cycle. In the absence of unacceptable toxicity or disease progression, treatment may continue for as long as tolerated.
  Interventions: Drug: Vismodegib

INTERVENTIONS:
Drug: Vismodegib
  Other Names: Erivedge

SUMMARY:
The purpose of this research study is to evaluate an investigational drug (Vismodegib) for Pontine Glioma that is growing or has come back (reoccurred). This study will look at the tumors response to the study drug, Vismodegib, and will also look at the safety and tolerability of Vismodegib.

Vismodegib has been tested in multiple adult clinical trials and one pediatric trial. Laboratory testing in pontine gliomas suggests that this drug may be effective in treating this disease.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have radiographically proven diffuse intrinsic pontine glioma and confirmation of residual disease after initial therapy or at the time of recurrence/progression as confirmed by MRI of the brain
* Subjects must be age ≥3 years and ≤ 18 years
* Diffuse intrinsic pontine glioma with measurable disease after receiving radiotherapy either concurrent with or followed by ≤ 2 prior courses of chemotherapy
* Measurable disease as defined by:

Measurable tumor >10mm by MRI

* Karnofsky performance status (PS) 60-100% (for patients > 16 years of age) OR Lansky PS 60-100% (for patients ≤ 16 years of age)
* Body surface area > 0.67 m2 and ≤ 2.21 m2
* Life expectancy of at least 2 months
* A negative urine pregnancy test is required for female participants of child bearing potential (≥13 years of age or after onset of menses)
* Acceptable liver function as defined by:

  1. Bilirubin ≤ 1.5 times upper limit of normal
  2. AST (SGOT), ALT (SGPT) and Alkaline phosphatase ≤ 2.5 times upper limit of normal
* Creatinine clearance or radioisotope GFR ≥ 70 mL/min OR serum creatinine based on age as follows:

  * 0.8 mg/dL (for patients ≤ 5 years of age)
  * 1.0 mg/dL (for patients 6 to 10 years of age)
  * 1.2 mg/dL (for patients 11 to 15 years of age)
  * 1.5 mg/dL (for patients > 15 years of age)
* Acceptable hematologic status as defined by:

  1. Granulocyte ≥ 1500 cells/mm3
  2. Platelet count ≥ 100,000 (plt/mm3)
  3. Serum albumin ≥ 2.5 g/dL
* Urinalysis:

  a. No clinically significant abnormalities
* Acceptable coagulation status as defined by:

  1. PT/INR less than 1.5
  2. PTT within normal limits
* Subjects must be able to swallow and retain oral medication
* Female post-pubertal study subjects need to agree to use one of the more effective birth control methods during treatment and for 7 (seven) months after treatment is stopped. These methods include total abstinence (no sex), oral contraceptives ("the pill"), an intrauterine device (IUD), levonorgestrol implants (Norplant), or medroxyprogesterone acetate injections (Depo-provera shots).
* Male post-pubertal study subjects need to agree to use condoms with spermicide, even after a vasectomy, during sexual intercourse with female partners while being treated with Erivedge capsule and for 2 months after the last dose to avoid exposing an embryo or fetus to Vismodegib.
* Voluntarily signed and dated a written IRB-approved informed consent by parent or legal guardian of subject

Exclusion Criteria:

* Concurrent anti-cancer therapy (chemotherapy, radiation therapy, surgery, immunotherapy, hormonal therapy, biologic therapy) other than the ones specified in the protocol. Patients must have discontinued the above cancer therapies for generally about 3 weeks (8 weeks for radiotherapy) prior to the first dose of study medication, as well as recovered from toxicity (to ≤ than grade 2 except for alopecia) induced by previous treatments.
* Currently receiving another investigational medicinal product.
* Uncontrolled concurrent illness including, but not limited to:

  1. Active, uncontrolled bacterial, viral, or fungal infections requiring systemic therapy
  2. Diarrhea of any cause ≥ CTCAE grade 2
  3. Psychiatric illness/social situations that would compromise patient safety or limit compliance with study requirements including maintenance of a compliance/pill diary
  4. Any kind of malabsorption syndrome significantly affecting gastrointestinal function
* Pregnant or nursing female patients. NOTE: If a female patient becomes pregnant or suspects that she is pregnant while participating in this study, she should stop taking study drug and immediately inform her treating physician immediately.
* Prior therapy with a Hedgehog inhibitor
* Unwillingness or inability to comply with procedures required in this protocol
* Serious nonmalignant disease (e.g., hydronephrosis, liver failure, or other conditions) that could compromise protocol objectives in the opinion of the investigator and/or the sponsor.
* History of Congestive Heart Failure (CHF) or ventricular arrhythmia requiring medication.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2013-05; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giselle Sholler, MD, Study Chair — Beat Childhood Cancer at Atrium Health; Albert Cornelius, MD, Principal Investigator — Helen DeVos Children's Hospital
Locations (2):
- United States (2):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Helen DeVos Children's Hospital, Grand Rapids, Michigan

REFERENCES:
- See also: Beat Childhood Cancer — https://beatcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Vismodegib: Vismodegib will be dosed at 150mg-300mg orally (max dose: 300mg) once a day on days 1 to 28 of a 28-day cycle. In the absence of unacceptable toxicity or disease progression, treatment may continue for as long as tolerated.
  Vismodegib
Period: Overall Study
Arm/Group | Vismodegib
Started | 9
Completed | 0
Not Completed | 9
Not completed — Lack of Efficacy | 4
Not completed — Physician Decision | 2
Not completed — Withdrawal by Subject | 2
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Vismodegib
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Days Participants Experienced Progression Free Survival (PFS)
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or the appearance of new lesions.
Time Frame: 5 years
Measure: Median (Full Range); unit: Days
Arm/Group | Vismodegib
Number analyzed (Participants) | 4
Days | 60 [20 to 143]

2. Secondary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability
Description: To determine the safety and tolerability of Vismodegib as a single agent in pediatric and young adult patients with refractory or recurrent pontine glioma
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Vismodegib
Number analyzed (Participants) | 9
participants | 4

3. Secondary Outcome: Determine the Median Overall Survival (OS) of Participants
Description: Overall Survival (OS) and clinical benefit (ORR + stable disease, SD)
Time Frame: 2 years
Population: Not evaluated due to early closure. Study data does not exist.
Arm/Group | Vismodegib
Number analyzed (Participants) | 0

4. Secondary Outcome: Evaluate the Impact of Quality of Life of Children Receiving Vismodegib Using PedsQL Questionnaires
Description: Evaluate the impact of Quality of Life of children receiving Vismodegib using PedsQL questionnaires
Time Frame: 2 years
Population: QOL's not collected due to early closure of study. Data not collected or analyzed threfore no data exists.
Arm/Group | Vismodegib
Number analyzed (Participants) | 0

5. Secondary Outcome: Determine the Response Rates of Participants Based on Activation (or no Activation) of Their Hedgehog Signaling Pathway
Description: To determine the objective response rates (partial and complete response) for patients without and with evidence of activation of Hedgehog signaling pathway in their tumors
Time Frame: 3 years
Population: No samples collected for hedgehog pathway. No data exists.
Arm/Group | Vismodegib
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: New adverse events collected from first dose of study drug to 30 days past last dose of study drug. Related adverse events followed until resolution.
Arm/Group | Vismodegib
Serious Adverse Events (participants affected / at risk) | 1/9
Other Adverse Events (participants affected / at risk) | 4/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vismodegib (N=9)
Choking event resulting in death (General disorders) | 1 (1) — Subject choked on a hot dog resulting in death. Unrelated to study.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vismodegib (N=9)
Alopecia (General disorders) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Gastoesophageal Reflux Disease (Gastrointestinal disorders) | 1 (1)
Increased GGT (Blood and lymphatic system disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No